CLINICAL TRIAL: NCT04283435
Title: Effect of Sildenafil on Uterine and Endometrial Vasculature in Women With Thin Endometrium Having Frozen-Thawed IVF Cycles
Brief Title: Endometrial Effects of Sildenafil in Frozen-Thawed Cycles in Women With Thin Endometrium
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Eman Elkattan, Associate professor, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: PROTOCOL 500
Record Dates: First submitted 2020-02-18; First posted 2020-02-25 (Actual); Last update posted 2021-08-20 (Actual); Status verified 2021-08

CONDITIONS: IVF; Endometrial Receptivity
MeSH Terms: interventions — Sildenafil Citrate; Estradiol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: One hundred envelopes will be numbered serially and in each envelope the corresponding letter which denotes the allocated group will be put according to randomization table. When the first patient arrives, the first envelope will be opened and the patient will be allocated according to the letter inside.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- estradiol valerate + placebo (Placebo Comparator): preparation of the endometrium with Estradiol valerate 2mg/day (every 8 hours)(white tablets of cycloprogenova) .from the first day of the cycle till 12th day and we add placebo from the first day of the cycle till the day of start progesterone (we stop 3 days before embryo transfer).
  Interventions: Other: Placebo; Drug: Estradiol Valerate
- estradiol valerate + Sildenafil citrate (Experimental): We add Sildenfil citrate 50 mg daily from the first day of the period till the day of starting the progesterone. and stop 3 days before the embryo transfer.
  Interventions: Drug: Sildenafil Citrate; Drug: Estradiol Valerate

INTERVENTIONS:
Drug: Sildenafil Citrate — Sildenafil Citrate 50 mg tablets taken from the first day of the cycle till the day we start progesterone (we stop 3 days before embryo transfer)
  Arms: estradiol valerate + Sildenafil citrate
Other: Placebo — Placebo tablet (multivitamins),Pregnacare vitamins (Vitabiotics,UK)
  Other Names: Pregnacare vitamins (Vitabiotics,UK)
  Arms: estradiol valerate + placebo
Drug: Estradiol Valerate — Estradiol valerate tablets 2mg every 8 hours daily starting from the fist day of the cycle till 12th day of the menstrual cycle.

SUMMARY:
Management of Thin endometrium in IVF is challenging. Thin endometrium is often defined as <7 mm or < 8 mm on the day of Human Gonadotropin administration(Bu and Sun, 2015; Wu et al., 2014).

Its incidence is 1-2.5% in most studies ( AlGhamdi et al.,2008).

Endometrial thickness and endometrial vascularity is closely linked to endometrial receptivity.Improving endometrial receptivity is a predictor of the success in IVF.

Many medications have been tried to improve endometrial thickness as Aspirin,sildenafil citrate,luteal estradiol and Granulocyte colony stimulating factor.

Nitric oxide (NO) is a key signaling molecule involved in the vasodilator response of smooth muscle cells. NO activates the cyclic guanosine monophosphate (cGMP)/protein kinase G (PKG) pathway within smooth muscle cells to promote smooth muscle cell relaxation. Sildenafil citrate inhibits phosphodiesterase 5 (PDE5) maintaining activation of cGMP and PKG and maximizing the effect of existing NO, thus facilitating smooth muscle cell relaxation. The potent vasodilator action of sildenafil has led researchers to evaluate sildenafil as a treatment in assisted reproduction where low uterine blood flow is perceived to be a contributor to implantation failure (Fairouzabadi et al.2013).

The investigators aim at this study to investigate the role of sildenafil citrate on endometrial and subendometrial vasculature in women with thin endometrium undergoing Frozen-Thawed IVF cycles.

DETAILED DESCRIPTION:
This is a Randomised-controlled trial .The investigators recruited 100 women who are known to have thin endometrium in previous IVF cycles (failed/cancelled cycles).

They are randomised into group A (50 women) : preparation of the endometrium with Estradiol valerate 2mg/day (every 8 hours)(white tablets of cycloprogenova,Payer,Germany) from the first day of the cycle till 12th day and The investigators add placebo from the first day of the cycle till the day of starting progesterone (It will be stopped 3 days before embryo transfer).Group B (50 women): The investigators add Sildenafil citrate (Viagra,pfizer,United states) to the estradiol valerate. Sildenafil 50 mg will be used daily from the first day of the cycle till the day of starting progesterone (It will be stopped 3 days before embryo transfer). The embryos will be transferred depending on their age on day 3 or day 5.

At the transfer date ,the investigators will assess the endometrial thickness, endometrial volume, uterine artery doppler indices (RI,PI) as well as 3D endometrial vascular indices (VI,FI,VFI) .

ELIGIBILITY:
Inclusion Criteria:

* Women (25 -40 years) undergoing IVF frozen-Thawed cycles and known to have good quality embryos.
* previous thin endometrium (< 8mm on at least 3 previous cycles) with normal Hysteroscopy findings

Exclusion Criteria:

* women less than 25 years old or more than 40 years old.
* abnormal hysteroscopic findings.
* women with congenital uterine anomalies.
* History of previous uterine surgery
* Any contraindication to Sildenafil as Previous history of cardiac disease or stroke.

Ages: 25 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Females undergoing IVF
Enrollment: 100 (Estimated)
Dates: Start 2021-09-01 (Estimated); Primary Completion 2022-03-01 (Estimated); Study Completion 2022-03-01 (Estimated)

PRIMARY OUTCOMES:
Clinical Pregnancy rate | 2 weeks after embryo transfer

SECONDARY OUTCOMES:
endometrial thickness | at the time of embryo transfer
Endometrial volume | at the time of embryo transfer
Uterine artery doppler indices | at the time of embryo transfer
3D endometrial and subendometrial vascular indices(VI,FI.VFI) | at the time of embryo transfer

CONTACTS AND LOCATIONS:
Locations (1):
- Cairo University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No